CLINICAL TRIAL: NCT04155814
Title: Bioequivalence Study Assessing a Single Dose of Iron Sucrose Injection (Baxter) or a Single Dose of Venofer® Injection in Healthy Adult Subjects
Brief Title: Bioequivalence Study Assessing Iron Sucrose or Venofer® in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BXU537298; QSC202208 (Other: Quotient)
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Bioequivalance
MeSH Terms: interventions — Ferric Oxide, Saccharated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Iron Sucrose Injection (Experimental): IV injection (5 mL), delivered over 5 minutes to subjects that have been fasted for a minimum of 10 hours.
  Interventions: Drug: Iron Sucrose Injection
- Venofer Injection (Active Comparator): IV injection (5 mL), delivered over 5 minutes to subjects that have been fasted for a minimum of 10 hours.
  Interventions: Drug: Venofer Injection

INTERVENTIONS:
Drug: Iron Sucrose Injection — USP 100 mg/5 mL (20 mg/mL), solution for IV injection, 100 mg unit dose strength
  Arms: Iron Sucrose Injection
Drug: Venofer Injection — (Iron Sucrose 20 mg/mL), solution for IV injection, 100 mg unit dose strength
  Arms: Venofer Injection

SUMMARY:
This study evaluates the bioequivalence, pharmacokinetic (PK) profile, and safety and tolerability of Iron Sucrose (Test Product) relative to that of Venofer® in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or non-pregnant, non-lactating healthy females
* Age 18 to 55 years of age (both inclusive)
* Must, in the opinion of the investigator, be in good health based upon medical history, physical examination (including vital signs and ECGs) and clinical laboratory tests assessed at the time of screening
* Body mass index (BMI) of 18.0 to 32.0 kg/m2 and a minimum body weight of 40 kg, or if outside the range, considered not clinically significant by the investigator
* Ferritin levels not less than the lower limit of normal as defined by clinical laboratory reference ranges for female and male subjects at screening only
* Transferrin Saturation (TSAT) not less than the lower limit of normal as defined by clinical laboratory reference ranges for female and male subjects at screening only
* Hemoglobin levels not less than the lower limit of normal as defined by clinical laboratory reference ranges for male and female subjects
* Must agree to use an adequate method of contraception:

  * For male subjects: Subjects willing to follow approved birth control methods (a double barrier method) for the duration of the study as judged by the investigator(s), such as condom with spermicide, condom with diaphragm, or abstinence. Subjects should also not donate sperm during this time.
  * For female subjects: Female subjects of childbearing potential, defined as a woman < 55 years of age who has not had a partial or full hysterectomy or oophorectomy, must have a negative urine pregnancy test at screening and a negative beta human chorionic gonadotropin (β-hCG) pregnancy test at admission. Subjects of childbearing potential must use a medically acceptable means of contraception during their participation in the study
* Non-smoker, defined as: Non-smoker for > 12 months (i.e., subject has not smoked or used any tobacco product, e-cigarettes, and nicotine replacement products for the 12 months prior to the start of the study) based on subject report.
* Must be willing and able to comply with all study requirements
* Must be able to understand a written informed consent, which must be obtained prior to initiation of study procedures

Exclusion Criteria:

* Hypersensitivity to iron sucrose or iron products
* Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hay fever is allowed unless it is active
* Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
* Clinically significant abnormal biochemistry, hematology or urinalysis as judged by the investigator
* History of iron deficiency within 6 months prior to screening
* History of anemia within 6 months prior to screening
* Suspicion of iron overload as evidenced by both elevated serum TSAT and serum ferritin levels
* History of hemochromatosis
* Bleeding disorders, acute bleeding or recently documented hemorrhage
* Females with history of hypermenorrhea or menorrhagia
* History of cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological or psychiatric disease or disorder, as judged by the investigator
* Must not have significant serious skin disease, including rash, food allergy, eczema, psoriasis, or urticaria
* Female subjects who are currently pregnant, lactating, or planning to become pregnant during the study period
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
* Positive drugs of abuse test result or history of drug abuse in the past 6 months based on subject report
* Positive urinalysis test for alcohol at screening or history of alcoholism in the past 6 months based on subject report
* Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 Units = 125 mL glass of wine, depending on type)
* Administration of an injectable drug within 14 days prior to drug administration in this study
* Subjects who are taking, or have taken, any prescribed or over-the-counter drug (other than up to 4 g per day acetaminophen in the 14 days before IMP administration, hormonal contraceptives, or hormone replacement therapy. Exceptions may apply on a case by case basis, if considered not to interfere with the objectives of the study, as agreed by the PI and sponsor's medical monitor
* Use of iron supplements (including iron-containing multivitamins) within 3 months of the first dose IMP administration in the study
* Have poor venous access that limits phlebotomy
* Subjects who have donated blood (1 unit = 450 mL) within 3 months prior to the first dose of the study drug and plasma within 7 days prior to the first dose of the study drug.
* Subjects who have received any IMP in a clinical research study within 5 half-lives or within 30 days prior to first dose. However, in no event, shall the time between last receipt of IMP and first dose be less than 30 days
* Subjects who are study site employees, or immediate family members of a study site or sponsor employee
* Subjects who have previously been enrolled in this study
* Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 196 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Cmax(delta) | Hours before injection (24, 12, 0.25); Minutes after end of injection (1, 5, 10, 15, 30, 45); Hours after end of injection (1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 16, 24, 36)
  Maximum concentration (Cmax) across all time points for the delta difference between Total Iron (TI) and Transferrin Bound Iron (TBI). This is a PK test parameter to compare bioequivalence of two drug products.
AUC0-t(delta) | Hours before injection (24, 12, 0.25); Minutes after end of injection (1, 5, 10, 15, 30, 45); Hours after end of injection (1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 16, 24, 36)
  Area under the concentration curve (AUC) from time zero to last time of quantifiable concentration (Tlast) for the delta difference in AUC0-t between TI and TBI. This is a PK test parameter to compare bioequivalence of two plasma drug products.

SECONDARY OUTCOMES:
Cmax | Hours before injection (24, 12, 0.25); Minutes after end of injection (1, 5, 10, 15, 30, 45); Hours after end of injection (1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 16, 24, 36)
  Maximum concentration (Cmax) across all time points for both TI and TBI. This is a PK test parameter to compare bioequivalence of two plasma drug products.
AUC0-t | Hours before injection (24, 12, 0.25); Minutes after end of injection (1, 5, 10, 15, 30, 45); Hours after end of injection (1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 16, 24, 36)
  Area under the concentration-time curve (AUC) from time zero to last sample time for both TI and TBI. This is a PK test parameter to compare bioequivalence of two drug products.
AUC0-inf | Hours before injection (24, 12, 0.25); Minutes after end of injection (1, 5, 10, 15, 30, 45); Hours after end of injection (1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 16, 24, 36)
  Area under the concentration-time curve (AUC) from time zero extrapolated to infinity for both TI and TBI. This is a PK test parameter to compare bioequivalence of two drug products.
Tmax | Hours before injection (24, 12, 0.25); Minutes after end of injection (1, 5, 10, 15, 30, 45); Hours after end of injection (1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 16, 24, 36)
  Time of occurrence of Cmax (Tmax) for both TI and TBI. This is a PK test parameter to compare bioequivalence of two drug products.
t1/2 | Hours before injection (24, 12, 0.25); Minutes after end of injection (1, 5, 10, 15, 30, 45); Hours after end of injection (1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 16, 24, 36)
  Terminal phase half-life (t1/2) for both TI and TBI. This is a PK test parameter to compare bioequivalence of two drug products.
Vz | Hours before injection (24, 12, 0.25); Minutes after end of injection (1, 5, 10, 15, 30, 45); Hours after end of injection (1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 16, 24, 36)
  Volume of distribution (Vz) for both TI and TBI. This is a PK test parameter to compare bioequivalence of two drug products.
CL | Hours before injection (24, 12, 0.25); Minutes after end of injection (1, 5, 10, 15, 30, 45); Hours after end of injection (1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 16, 24, 36)
  Total body clearance (CL) for extravascular administration calculated by Dose/AUC for both TI and TBI. This is a PK test parameter to compare bioequivalence of two drug products.
Percentage of AUCex | Hours before injection (24, 12, 0.25); Minutes after end of injection (1, 5, 10, 15, 30, 45); Hours after end of injection (1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 16, 24, 36)
  AUC0-inf due to extrapolation (AUCex) from Tlast to infinity calculated by: 100 × (AUC0-inf-AUC0-t)/AUC0-inf (%AUCex) for both TI and TBI. This is a PK test parameter to compare bioequivalence of two drug products.
Number of participants with clinically significant laboratory abnormalities | Day -28 (Screening) through Day 10 (Follow-up)
  Any clinically significant abnormality will also be reported as an AE.
Number of participants with clinically significant findings on physical examinations | Day -28 (Screening) through Day 10 (Follow-up)
  Any clinically significant abnormality will also be reported as an AE.
Number of participants with clinically significant changes to ECG parameters | Day -28 (Screening), Day -2, 0.25 hours before injection, and 6, 24 and 36 hours after end of injection
  Any clinically significant abnormality will also be reported as an AE.
Number of participants with occurrence of adverse events (AEs) | Day -28 (Screening) through Day 30
  An AE is any untoward medical occurrence in a subject that occurs either before dosing (referred to as a pre-dose AE) or once a medicinal product has been administered, including occurrences which are not necessarily caused by or related to that product.
Number of participants with occurrence of adverse events of special interest | Day -28 (Screening) through Day 30
  Special interest items includes hypersensitivity reactions including anaphylactic/anaphylactoid reactions.

CONTACTS AND LOCATIONS:
Locations (1):
- Baxter Investigational Site, Miami, Florida, United States